CLINICAL TRIAL: NCT05796622
Title: A Randomized Controlled Trial Evaluating an Innovative HIV Self-testing Service With Online Real-time Instruction, Pre-test and Post-test Counselling Provided by a Fully-automated Artificial Intelligence Chatbot (HIVST-Chatbot)
Brief Title: Evaluating an Innovative HIV Self-testing Service With Counseling Provided by a Chatbot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MSS349R
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Behaviors, Health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIVST-Chatbot (HIV self-testing services with counseling provided by a Chatbot) (Experimental): Promote and implement HIV self-testing (HIVST) services with real-time counselling provided by a fully-automated artificial intelligence Chatbot (HIVST-Chatbot)
  Interventions: Behavioral: HIVST-Chatbot (HIV self-testing services with counseling provided by a Chatbot)
- HIVST-OIC (HIV self-testing services with counseling provided by administrators) (Active Comparator): Promote and implement HIV self-testing (HIVST) services with real-time counselling provided by trained administrators)
  Interventions: Behavioral: HIVST-OIC (HIV self-testing services with counseling provided by administrators)

INTERVENTIONS:
Behavioral: HIVST-Chatbot (HIV self-testing services with counseling provided by a Chatbot) — Promote and implement HIVST-Chatbot
  Arms: HIVST-Chatbot (HIV self-testing services with counseling provided by a Chatbot)
Behavioral: HIVST-OIC (HIV self-testing services with counseling provided by administrators) — Promote and implement HIVST-OIC
  Arms: HIVST-OIC (HIV self-testing services with counseling provided by administrators)

SUMMARY:
A parallel-group non-inferiority randomized controlled trial will then be conducted to evaluate the performance of HIVST-Chatbot. A total of 528 Hong Kong Chinese speaking men who have sex with men (MSM) aged ≥18 years who have access to live-chat applications are recruited from multiple sources. Those who are diagnosed as HIV positive are excluded. Participants are 1:1 randomized into the intervention group (n=264) or the control group (n=264). The research team will implement the HIVST-Chatbot (HIVST services with real-time counselling provided by a fully-automated artificial intelligence Chatbot) in the intervention group and HIVST-OIC (HIVST with real-time counselling provided by trained administrators) in the control group. Participants completed two telephone surveys at baseline and six months afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese-speaking men aged at least 18 years old
* Having had anal intercourse with at least one man in the past six months
* Willing to leave contact information and be followed up at Month 6
* Having access to the online live-chat application (WhatsApp)
* Not intending to leave Hong Kong for one month consecutively within the next six months

Exclusion Criteria:

* Self-reported as HIV positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male at birth
Enrollment: 564 (Estimated)
Dates: Start 2023-04-16 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Uptake of HIV self-testing | 6 months
  Proportion of participants who use HIV self-testing during the 6-month follow-up period
Proportion of HIV self-testing users receiving counselling along with testing | 6 months
  Proportion of HIV self-testing users receiving counselling along with testing during the 6-month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen S, Yu FY, Fang Y, Yau J, Ng N, Zhang Q, Ni Z, Duong MC, Sun F, Mo PKH, Wang Z. Chatbot-Delivered Real-Time Support to Improve HIV Self-Testing Rates: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2544821. doi: 10.1001/jamanetworkopen.2025.44821. PMID 41284298
- [Derived] Chen S, Zhang Q, Chan CK, Yu FY, Chidgey A, Fang Y, Mo PKH, Wang Z. Evaluating an Innovative HIV Self-Testing Service With Web-Based, Real-Time Counseling Provided by an Artificial Intelligence Chatbot (HIVST-Chatbot) in Increasing HIV Self-Testing Use Among Chinese Men Who Have Sex With Men: Protocol for a Noninferiority Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 30;12:e48447. doi: 10.2196/48447. PMID 37389935